CLINICAL TRIAL: NCT04635150
Title: National Evaluation of the Close Collaboration With Parents Training. Enhancing Parents' Presence and Participation During Neonatal Intensive Care.
Brief Title: National Evaluation of the Close Collaboration With Parents Training
Acronym: VVME5
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Turku University Hospital (Other Government)
Collaborators: University of Turku (Other)
Responsible Party: Principal Investigator, Liisa Lehtonen, Professor, Turku University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: K37/12
Record Dates: First submitted 2020-11-12; First posted 2020-11-18 (Actual); Last update posted 2020-11-18 (Actual); Status verified 2020-11

CONDITIONS: Parent-Child Relations; Parenting; Infant, Newborn, Disease
Keywords: NICU; Family centered care; Parent-infant closeness; Skin-to-skin
MeSH Terms: conditions — Disease

STUDY DESIGN:
Intervention Model Description: Pre-post intervention study with different cohorts before and after the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Post-intervention parents and staff (Experimental): An educational intervention for the multidisciplinary staff of a neonatal intensive care unit.
  Interventions: Behavioral: Close Collaboration with Parents

INTERVENTIONS:
Behavioral: Close Collaboration with Parents — Close Collaboration with Parents Training Program is an educational intervention for multidisciplinary NICU staff initially developed and implemented at Turku University Hospital to promote FCC. The intervention consists of four phases lasting 4 to 5 months each. First the healthcare staff learn to observe infant behavior. This phase aims at identifying the individual needs and features of each infant. After that, the staff observe infant behavior with the parents and learn to actively listen to parents' perceptions about their infant. During the phase III, staff learn to know the individual story of the family and their infant, which supports partnership between staff and parents. Finally, staff learn to integrate parents in decision-making and collaboratively plan the transition to home. The training is delivered through facilitator-network model in which local mentors are trained by the trainer mentors and supervisors.

SUMMARY:
The aim of this study was to evaluate the effects of an educational intervention for neonatal staff on parent-infant physical closeness during their infant's stay in the Neonatal Intensive Care Unit (NICU) and parents' and staff perception on family centered care in the unit. This pre-post intervention study was carried out in nine hospitals in Finland in 2012 through 2018. Data was collected by using daily parental diaries, daily text message questions to parents and an audit interview for the staff.

DETAILED DESCRIPTION:
The aim of this study was to evaluate the effects of an educational intervention for neonatal staff on parent-infant physical closeness during their infant's stay in the Neonatal Intensive Care Unit (NICU) and parents' and staff perception on family centered care (FCC) in the unit. We hypothesized that parents spend more time in the unit and have more skin-to skin contact with their infant after the intervention compared to the time before the intervention. We also hypothesized that care culture becomes more family centered after the intervention both from parent and staff perspectives.

Study NICUs and participants This study was an intervention study, comparing the situation before and after the intervention. It was carried out in nine NICUs in Finland, including two level III hospitals and seven level II hospitals. The study progressed stepwise between May 2012 and September 2018; two or three hospitals participated in the study simultaneously. The study permission was granted by the Hospital District of Southwest Finland (T57/2012) and separately by each study site.

The study participants were recruited during three-month periods before and after the Close Collaboration with Parents training program, which lasted for 18 months. Every parent of an infant estimated to stay in the NICU longer than three days was approached. Other inclusion criteria were: 1) the infant had no major congenital anomalies or syndromes, 2) the parents spoke Finnish or Swedish, 3) the family lived in the catchment area of the hospital. A log including infant's gestational age, birth weight, the length of hospital period and the distance to home was kept for all admissions of infants with a length of stay longer than 3 days to identify eligible parents and evaluate drop-out rate.

The staff introduced the study protocol to parents and gave them at least one day to consider their participation. After the parents signed the informed consent form, they were given instructions for use of the closeness diaries and text messages. The parents provided infant characteristics (including gestational age, birthweight, birth head circumference, sex, mode of delivery, and whether the infant was a singleton/multiple or had siblings) and family characteristics (including parents' age, education, socio-economic status and the distance from the hospital to home).

Closeness diary The duration of parents' presence in the NICU and skin-to-skin contact (SSC) was reported with closeness diaries. Presence in the unit was defined by being inside the unit, not necessarily all the time in the room of the baby. SSC was defined as the baby lying on the parent's bare chest dressed only in a diaper and a cap if necessary. On the diary, there were four different timelines where parents filled in the time spent in NICU and SSC with their infant: mother present, mother SSC, father present, and father SSC. Parents were asked to fill in the diaries from the time of recruitment until discharge. During data collection, the diaries were stored in a folder at the bedside so that other families or nurses did not see the diaries.

Intervention The Close Collaboration with Parents intervention was developed based on theoretical evidence from infant neurobehavioral and attachment theories. The training is based on a multi-method learning philosophy using theoretical teaching, hands-on teaching at bedside, and reflective discussions supporting simultaneous implementation of practice change. The intervention teaches new skills to the entire staff of a unit to collaborate with parents in order to support parents' presence and involvement in infant's care. The original intervention was condensed to a structured 18-month-long training including four phases. A facilitator network model was used including local mentors trained by the trainer mentors and a supervisor.

BLISS Audit tool The data from staff were collected using the Bliss Baby Charter Audit Tool with permission of Bliss organization. The audit tool is a self-assessment instrument identifying areas of improvement in the quality of FCC in NICUs. The tool has 141 statements divided into seven core principles which summarize the care, respect and support that infants and their parents should receive. All seven principles contain different categories of family-centered care (as defined by Bliss). The categories are 1) Active care by parent and staff, (18 criteria), 2) Parent and family support (17 criteria), 3) Communication (6 criteria), 4) Developmental care (9 criteria), 5) Empowered decision making (10 criteria), 6) Facilities (17 criteria) ,7) Guidelines and policies (17 criteria), 8) Staff skills and training (12 criteria), 9) Information provision (27 criteria) and 10) Service improvement and parent involvement (8 criteria).

DigiFCC Parents evaluated the quality of FCC with DigiFCC-P tool by answering to the text-message questions delivered by mobile phones. The tool was developed for the evaluation of the Close Collaboration with Parents training Program. Parents received one randomized question from seven questions every evening during their infant hospitalization. The tool was further developed based on feedback from parents, staff, and researchers to improve its content validity and feasibility after the first four hospitals. In hospitals 5 to 9, parents received one randomized question from nine questions every evening during their infant hospitalization. The questions were: 1) To what extent did the staff listen to you today? 2) To what extent did you participate in your baby's care today? 3) To what extent did the guidance provided by the staff meet your needs today? 4) To what extent was your opinion considered in decisions made about your baby today? 5) To what extent did you trust the staff in the care of your baby today? 6) To what extent did the staff trust you in the care of your baby today? 7) To what extent did you participate in the discussion during the medical round? 8) To what extent did the information provided by the staff meet your needs today? 9) To what extent did the staff offer you emotional support today? Parents rated their responses on a 5-point Likert scale in hospitals 1 to 4, and in a 7-point Likert scale in hospitals 5 to 9 (1-7, with 1= not at all, 7= very much) or 0, if they were not in the NICU that day.

Nurses evaluated the quality of FCC with the DigiFCC-N tool. Nurses answered corresponding questions with the parents' questions exception of the question that concerned parental participation in the medical round. Questions to nurses were in a form: "To what extent did you listen to parents today?" Nurses gave the answer through a Web questionnaire using the computer assigned for the research purpose. Nurses replied one randomized question after each work shift during a 3-months study period before and after the training program.

Statistical methods Parents' presence was defined as at least one parent present. Mothers' and fathers' presence and SSC were also analysed separately. We compared the pre-intervention and post-intervention cohorts adjusting for gestational age, siblings in the family, and the neonatal unit in the statistical model. These confounders were chosen based their significance on parents' presence. The comparison of presence and SSC was analyzed using a linear model, where cohorts were independent families, siblings in the family and neonatal unit were handled as categorical variables, and gestational age as a continuous covariate. Analyses were performed for mother and father separately and then also as combined (at least one parent present, either parent SSC). All diaries until the last one were included in the analyses, also the days without presence or SSC or missing data. All statistical tests were performed as two-sided, with a significance level set at 0.05. The analyses were performed using SAS System, version 9.4 for Windows (SAS Institute Inc., Cary, NC, USA).

ELIGIBILITY:
1. Parents

   Inclusion Criteria for parents:
   * Every parent of an infant estimated to stay in the NICU longer than three days was approached.

   Exclusion Criteria:
   * Infant had major congenital anomalies or syndromes,
   * Parents spoke neither Finnish or Swedish,
   * Family lived outside the catchment area of the hospital.
2. All staff members working at bedside and leadership.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 768 (Actual)
Dates: Start 2012-05-30 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Parental Closeness Diary of parents' presence | During the time the infant was cared for in the neonatal unit (up to 3 months), applicable to both cohorts of infants: those recruited before and after the intervention.
  Daily Closeness Diary including space for both mothers and fathers to indicate their presence in the neonatal unit (minutes/per day in 5-minute accuracy) to be filled in during all hospital days of the infant (up to 3 months).
Parental Closeness Diary of parent-infant skin-to-skin contact | During the time the infant was cared for in the neonatal unit (up to 3 months), applicable to both cohorts of infants: those recruited before and after the intervention. .
  Daily Closeness Diary including space for both mothers and fathers to indicate skin-to-skin contact with their infant (minutes/per day in 5-minute accuracy) to be filled in during all hospital days of the infant (up to 3 months). Skin-to-skin contact is defined as the infant is lying naked on a parent's chest.
Daily text message questions to both mothers and fathers/partners about parents' satisfaction to family centered care | During the time the infant was cared for in the neonatal unit (up to 3 months), applicable to both cohorts of infants: those recruited before and after the intervention.
  Both parents received one question (randomly out of 9 questions) every evening at 9 pm to report their satisfaction about the specific issue during that day.
Web questions for the staff about the quality of family centered care they have provided during their work shift | Three months before and three months after the intervention.
  Each staff member responded to one web question (randomly out of 8 questions) after each workshift about the quality of family centered care they had provided that day.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] He FB, Axelin A, Ahlqvist-Bjorkroth S, Raiskila S, Loyttyniemi E, Lehtonen L. Effectiveness of the Close Collaboration with Parents intervention on parent-infant closeness in NICU. BMC Pediatr. 2021 Jan 11;21(1):28. doi: 10.1186/s12887-020-02474-2. PMID 33430816